CLINICAL TRIAL: NCT06991465
Title: Organ Preservation in Rectal Adenocarcinoma Using Hypofractionated Pelvic Radiotherapy (Hypo-OPRA): A Phase II Clinical Trial
Brief Title: Organ Preservation in Rectal AdenoCa Using Hypofractionated Pelvic RT(Hypo-OPRA)
Acronym: Hypo-OPRA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neil Kopek (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor-Investigator, Neil Kopek, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-9472
Record Dates: First submitted 2025-05-12; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiotherapy; Folfox protocol; Capecitabine

STUDY DESIGN:
Intervention Model Description: To achieve a complete clinical response (cCR) to their preoperative treatment which opens the possibility of avoiding surgery and consequently preserving the rectum. There now exists a growing body of data from centres around the world validating the safety of a surveillance approach in clinical complete responders treated with LCCRT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated Pelvic Radiotherapy (Experimental): A single arm consisting of hypofractionated RT dose of 25 Gy in 5 fractions once daily fractions of intensity modulated radiotherapy (IMRT) with a simultaneous integrated boost up to 35 Gy on sites of gross disease (tumour and lymphadenopathy).
  Interventions: Radiation: Radiation Therapy; Drug: FOLFOX regimen; Drug: Capecitabine

INTERVENTIONS:
Radiation: Radiation Therapy — High Dose Hypofractionated Radiotherapy 35 Gy over 5 fractions.
  Other Names: Hyofractionated Radiotherapy
Drug: FOLFOX regimen — Radiosensitizing chemotherapy
Drug: Capecitabine — Radiosensitizing chemotherapy

SUMMARY:
The combination of preoperative pelvic RT - either long-course chemoradiotherapy (LCCRT) or short-course radiotherapy (SCRT)- followed by surgery has been the standard of care in the curative treatment of locally advanced adenocarcinoma of the rectum for decades. Some patients however achieve a complete clinical response (cCR) to their preoperative treatment which opens the possibility of avoiding surgery and consequently preserving the rectum. There now exists a growing body of data from centres around the world validating the safety of a surveillance approach in clinical complete responders treated with LCCRT.

DETAILED DESCRIPTION:
At McGill, SCRT is used routinely as a pre-operative radiotherapy schedule for locally advanced adenocarcinomas of the rectum. Likewise SCRT followed by chemotherapy is already used routinely at McGill as a pre-operative regimen for locally advanced rectal cancer with high risk features. Compelling registry data from Scandinavia shows that enduring clinical complete responses can be achieved after SCRT. To date, however, nearly all of the published data supporting a surveillance strategy in complete clinical responders is based on LCCRT. The present study proposes to explore further the organ preservation potential of SCRT.

Adopting a non-operative strategy in rectal cancer patients who achieve complete tumour regression avoids the risks of surgical morbidity and mortality, notably a sparing of the rectal sphincter muscles in the case of low-lying tumours and consequently avoidance of a permanent stoma.

Although multiple phase III trials support the routine use of SCRT in the pre-operative setting for locally advanced rectal adenocarcinoma, to date nearly all of the published data supporting a surveillance strategy in complete clinical responders is based on LCCRT. Compelling registry data from Scandinavia does show that enduring clinical complete responses can be achieved after short-course pelvic radiotherapy. Furthermore, the Rectal Cancer and Pre-operative Induction Therapy Followed by Dedicated Operation (RAPIDO) study demonstrated that, compared with LCCRT, SCRT followed by chemotherapy (SCRT-CH) has a higher pathologic complete response rate (29% versus 14%), less disease-related treatment failure, and superior distant metastasis-free survival.

Short-course pelvic radiotherapy with or without sequential chemotherapy can induce enduring clinical complete responders and the use of SCRT as part of a non-operative organ preservation strategy merits further prospective exploration. At McGill, SCRT is already used routinely as a pre-operative dose schedule for clinically node negative/N1 locally advanced adenocarcinomas of the rectum where downsizing is not required to achieve a sphincter sparing R0 resection. Likewise, since the publication of the RAPIDO trial, SCRT followed by FOLFOX/CAPOX chemotherapy has emerged as the preferred regimen at McGill for patients with high risk features (cT4 disease, cN2 and/or extramesorectal nodes, EMVI+, threatened or involved mesorectal fascia and/or sphincter muscles). The present phase II prospective study proposes to explore further the organ preservation potential of SCRT combined with a simultaneous integrated boost on sites of gross disease..

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive adenocarcinoma of the rectum
* Pelvic MRI defined disease (at least one of the following):

mesorectum involved or breached - includes involvement of adjacent organ(s) (T3-T4)

* Patients are considered medically fit for oncologic resection
* ECOG performance status 0 or 1
* No evidence of established metastatic disease (CT chest and abdomen)
* Absolute neutrophil count >1.5x109/L; platelets >100x109/L,
* Serum transaminase <3 x ULN;
* Adequate renal function (Cockroft Gault estimation >50 mL/min)
* Bilirubin <1.5 x ULN
* Ability to comply with oral medication
* Willingness and ability to give informed consent and comply with treatment and follow up schedule
* Age 18 or over

Exclusion Criteria:

* Previous chemotherapy
* Previous radiotherapy to the pelvis (including brachytherapy)
* Uncontrolled cardiorespiratory comorbidity (includes patients with inadequately controlled angina or myocardial infarction within 6 months of randomisation)
* T1 or T2 N0 disease without extra-mural venous invasion
* Unequivocal evidence of metastatic disease (includes resectable metastases)
* Major impairment of bowel function without defunctioning stoma/ileostomy (baseline grade 3 diarrhoea or clinically significant faecal incontinence
* Known dihydropyrimidine dehydrogenase deficiency
* History of another malignancy within the last 5 years except successfully treated basal cell cancer of skin or carcinoma in situ of uterine cervix.
* Known Gilberts disease (hyperbilirubinaemia)
* Taking warfarin or phenytoin or sorivudine
* Gastrointestinal disorder which would interfere with oral therapy and its bioavailability
* Pregnant, lactating, or pre-menopausal women not using adequate contraception
* Unfit to receive any study treatment or subsequent surgical resection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Hypo-fractionated Approach in 5 fractions for a dose of 35Gy | One year
  Rate of failure to achieve CR or the rate of recurrence after achieving CR

CONTACTS AND LOCATIONS:
Overall Officials: Neil Kopek, M.D., Principal Investigator — Radiation Oncologist - Radiation Oncology
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim H, Pedersen K, Olsen JR, Mutch MG, Chin RI, Glasgow SC, Wise PE, Silviera ML, Tan BR, Wang-Gillam A, Lim KH, Suresh R, Amin M, Huang Y, Henke LE, Park H, Ciorba MA, Badiyan S, Parikh PJ, Roach MC, Hunt SR. Nonoperative Rectal Cancer Management With Short-Course Radiation Followed by Chemotherapy: A Nonrandomized Control Trial. Clin Colorectal Cancer. 2021 Sep;20(3):e185-e193. doi: 10.1016/j.clcc.2021.03.003. Epub 2021 Apr 7. PMID 34001462
- [Result] Bahadoer RR, Dijkstra EA, van Etten B, Marijnen CAM, Putter H, Kranenbarg EM, Roodvoets AGH, Nagtegaal ID, Beets-Tan RGH, Blomqvist LK, Fokstuen T, Ten Tije AJ, Capdevila J, Hendriks MP, Edhemovic I, Cervantes A, Nilsson PJ, Glimelius B, van de Velde CJH, Hospers GAP; RAPIDO collaborative investigators. Short-course radiotherapy followed by chemotherapy before total mesorectal excision (TME) versus preoperative chemoradiotherapy, TME, and optional adjuvant chemotherapy in locally advanced rectal cancer (RAPIDO): a randomised, open-label, phase 3 trial. Lancet Oncol. 2021 Jan;22(1):29-42. doi: 10.1016/S1470-2045(20)30555-6. Epub 2020 Dec 7. PMID 33301740
- [Result] Nilsson PJ, Ahlberg M, Kordnejad S, Holm T, Martling A. Organ preservation following short-course radiotherapy for rectal cancer. BJS Open. 2021 Sep 6;5(5):zrab093. doi: 10.1093/bjsopen/zrab093. PMID 34686879
- [Result] Temple LK, Bacik J, Savatta SG, Gottesman L, Paty PB, Weiser MR, Guillem JG, Minsky BD, Kalman M, Thaler HT, Schrag D, Wong WD. The development of a validated instrument to evaluate bowel function after sphincter-preserving surgery for rectal cancer. Dis Colon Rectum. 2005 Jul;48(7):1353-65. doi: 10.1007/s10350-004-0942-z. PMID 15868235
- [Result] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Result] Appelt AL, Ploen J, Harling H, Jensen FS, Jensen LH, Jorgensen JC, Lindebjerg J, Rafaelsen SR, Jakobsen A. High-dose chemoradiotherapy and watchful waiting for distal rectal cancer: a prospective observational study. Lancet Oncol. 2015 Aug;16(8):919-27. doi: 10.1016/S1470-2045(15)00120-5. Epub 2015 Jul 5. PMID 26156652
- [Result] Glynne-Jones R, Hughes R. Critical appraisal of the 'wait and see' approach in rectal cancer for clinical complete responders after chemoradiation. Br J Surg. 2012 Jul;99(7):897-909. doi: 10.1002/bjs.8732. Epub 2012 Apr 27. PMID 22539154
- [Result] Maas M, Beets-Tan RG, Lambregts DM, Lammering G, Nelemans PJ, Engelen SM, van Dam RM, Jansen RL, Sosef M, Leijtens JW, Hulsewe KW, Buijsen J, Beets GL. Wait-and-see policy for clinical complete responders after chemoradiation for rectal cancer. J Clin Oncol. 2011 Dec 10;29(35):4633-40. doi: 10.1200/JCO.2011.37.7176. Epub 2011 Nov 7. PMID 22067400
- [Result] Dalton RS, Velineni R, Osborne ME, Thomas R, Harries S, Gee AS, Daniels IR. A single-centre experience of chemoradiotherapy for rectal cancer: is there potential for nonoperative management? Colorectal Dis. 2012 May;14(5):567-71. doi: 10.1111/j.1463-1318.2011.02752.x. PMID 21831177
- [Result] Habr-Gama A. Assessment and management of the complete clinical response of rectal cancer to chemoradiotherapy. Colorectal Dis. 2006 Sep;8 Suppl 3:21-4. doi: 10.1111/j.1463-1318.2006.01066.x. PMID 16813588
- [Result] Habr-Gama A, de Souza PM, Ribeiro U Jr, Nadalin W, Gansl R, Sousa AH Jr, Campos FG, Gama-Rodrigues J. Low rectal cancer: impact of radiation and chemotherapy on surgical treatment. Dis Colon Rectum. 1998 Sep;41(9):1087-96. doi: 10.1007/BF02239429. PMID 9749491
- [Result] Habr-Gama A, Gama-Rodrigues J, Sao Juliao GP, Proscurshim I, Sabbagh C, Lynn PB, Perez RO. Local recurrence after complete clinical response and watch and wait in rectal cancer after neoadjuvant chemoradiation: impact of salvage therapy on local disease control. Int J Radiat Oncol Biol Phys. 2014 Mar 15;88(4):822-8. doi: 10.1016/j.ijrobp.2013.12.012. Epub 2014 Feb 1. PMID 24495589
- [Result] Habr-Gama A, Perez RO, Nadalin W, Nahas SC, Ribeiro U Jr, Silva E Sousa AH Jr, Campos FG, Kiss DR, Gama-Rodrigues J. Long-term results of preoperative chemoradiation for distal rectal cancer correlation between final stage and survival. J Gastrointest Surg. 2005 Jan;9(1):90-9; discussion 99-101. doi: 10.1016/j.gassur.2004.10.010. PMID 15623449
- [Result] Habr-Gama A, Perez RO, Nadalin W, Sabbaga J, Ribeiro U Jr, Silva e Sousa AH Jr, Campos FG, Kiss DR, Gama-Rodrigues J. Operative versus nonoperative treatment for stage 0 distal rectal cancer following chemoradiation therapy: long-term results. Ann Surg. 2004 Oct;240(4):711-7; discussion 717-8. doi: 10.1097/01.sla.0000141194.27992.32. PMID 15383798
- [Result] Habr-Gama A, Perez RO, Proscurshim I, Campos FG, Nadalin W, Kiss D, Gama-Rodrigues J. Patterns of failure and survival for nonoperative treatment of stage c0 distal rectal cancer following neoadjuvant chemoradiation therapy. J Gastrointest Surg. 2006 Dec;10(10):1319-28; discussion 1328-9. doi: 10.1016/j.gassur.2006.09.005. PMID 17175450
- [Result] Maas M, Nelemans PJ, Valentini V, Das P, Rodel C, Kuo LJ, Calvo FA, Garcia-Aguilar J, Glynne-Jones R, Haustermans K, Mohiuddin M, Pucciarelli S, Small W Jr, Suarez J, Theodoropoulos G, Biondo S, Beets-Tan RG, Beets GL. Long-term outcome in patients with a pathological complete response after chemoradiation for rectal cancer: a pooled analysis of individual patient data. Lancet Oncol. 2010 Sep;11(9):835-44. doi: 10.1016/S1470-2045(10)70172-8. Epub 2010 Aug 6. PMID 20692872
- [Result] Hartley A, Ho KF, McConkey C, Geh JI. Pathological complete response following pre-operative chemoradiotherapy in rectal cancer: analysis of phase II/III trials. Br J Radiol. 2005 Oct;78(934):934-8. doi: 10.1259/bjr/86650067. PMID 16177017
- [Result] Gervaz PA, Wexner SD, Pemberton JH. Pelvic radiation and anorectal function: introducing the concept of sphincter-preserving radiation therapy. J Am Coll Surg. 2002 Sep;195(3):387-94. doi: 10.1016/s1072-7515(02)01308-x. No abstract available. PMID 12229948
- [Result] Bujko K, Nowacki MP, Nasierowska-Guttmejer A, Michalski W, Bebenek M, Kryj M. Long-term results of a randomized trial comparing preoperative short-course radiotherapy with preoperative conventionally fractionated chemoradiation for rectal cancer. Br J Surg. 2006 Oct;93(10):1215-23. doi: 10.1002/bjs.5506. PMID 16983741
- [Result] Rutten HJ, den Dulk M, Lemmens VE, van de Velde CJ, Marijnen CA. Controversies of total mesorectal excision for rectal cancer in elderly patients. Lancet Oncol. 2008 May;9(5):494-501. doi: 10.1016/S1470-2045(08)70129-3. PMID 18452860
- [Result] Paun BC, Cassie S, MacLean AR, Dixon E, Buie WD. Postoperative complications following surgery for rectal cancer. Ann Surg. 2010 May;251(5):807-18. doi: 10.1097/SLA.0b013e3181dae4ed. PMID 20395841
- [Result] Borowski DW, Bradburn DM, Mills SJ, Bharathan B, Wilson RG, Ratcliffe AA, Kelly SB; Northern Region Colorectal Cancer Audit Group (NORCCAG). Volume-outcome analysis of colorectal cancer-related outcomes. Br J Surg. 2010 Sep;97(9):1416-30. doi: 10.1002/bjs.7111. PMID 20632311
- [Result] van Gijn W, Marijnen CA, Nagtegaal ID, Kranenbarg EM, Putter H, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer: 12-year follow-up of the multicentre, randomised controlled TME trial. Lancet Oncol. 2011 Jun;12(6):575-82. doi: 10.1016/S1470-2045(11)70097-3. Epub 2011 May 17. PMID 21596621
- [Result] Sebag-Montefiore D, Stephens RJ, Steele R, Monson J, Grieve R, Khanna S, Quirke P, Couture J, de Metz C, Myint AS, Bessell E, Griffiths G, Thompson LC, Parmar M. Preoperative radiotherapy versus selective postoperative chemoradiotherapy in patients with rectal cancer (MRC CR07 and NCIC-CTG C016): a multicentre, randomised trial. Lancet. 2009 Mar 7;373(9666):811-20. doi: 10.1016/S0140-6736(09)60484-0. PMID 19269519
- [Result] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Result] Peeters KC, Marijnen CA, Nagtegaal ID, Kranenbarg EK, Putter H, Wiggers T, Rutten H, Pahlman L, Glimelius B, Leer JW, van de Velde CJ; Dutch Colorectal Cancer Group. The TME trial after a median follow-up of 6 years: increased local control but no survival benefit in irradiated patients with resectable rectal carcinoma. Ann Surg. 2007 Nov;246(5):693-701. doi: 10.1097/01.sla.0000257358.56863.ce. PMID 17968156
- [Result] Bosset JF, Collette L, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Ollier JC; EORTC Radiotherapy Group Trial 22921. Chemotherapy with preoperative radiotherapy in rectal cancer. N Engl J Med. 2006 Sep 14;355(11):1114-23. doi: 10.1056/NEJMoa060829. PMID 16971718
- [Result] Gerard JP, Conroy T, Bonnetain F, Bouche O, Chapet O, Closon-Dejardin MT, Untereiner M, Leduc B, Francois E, Maurel J, Seitz JF, Buecher B, Mackiewicz R, Ducreux M, Bedenne L. Preoperative radiotherapy with or without concurrent fluorouracil and leucovorin in T3-4 rectal cancers: results of FFCD 9203. J Clin Oncol. 2006 Oct 1;24(28):4620-5. doi: 10.1200/JCO.2006.06.7629. PMID 17008704